CLINICAL TRIAL: NCT03731325
Title: The Effect of Episodic Future Thinking on Weight-Loss
Brief Title: Episodic Future Thinking and Weight-Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Leonard Epstein, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201807151; R01HD080292 (NIH)
Record Dates: First submitted 2018-10-30; First posted 2018-11-06 (Actual); Results first posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-09

CONDITIONS: Overweight and Obesity
Keywords: Episodic future thinking; Obesity; Family based treatment
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Non-concurrent multiple baseline design;participants will be randomized to a 7 week, or 10 week group with staggered baseline periods followed by 4-8 weeks of the intervention consisting of FBT and EFT. Enrollment is for parent-child dyads.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Episodic Future Thinking Group 7-week baseline (Experimental): The experimental group will receive the Episodic Future Thinking (EFT) intervention after a 7-week baseline. EFT teaches individuals to pre-experience events, or think prospectively, about future events as if they were happening now [Atance].
  Interventions: Behavioral: Episodic Future Thinking Group
- Episodic Future Thinking Group 10-week baseline (Experimental): The experimental group will receive the Episodic Future Thinking (EFT) intervention after a 10-week baseline. EFT teaches individuals to pre-experience events, or think prospectively, about future events as if they were happening now [Atance].
  Interventions: Behavioral: Episodic Future Thinking Group

INTERVENTIONS:
Behavioral: Episodic Future Thinking Group — Participants in the Episodic Future Thinking (EFT) Group will train with EFT throughout the entire study. As part of the training, research staff will help participants create "cues." Cues are descriptions of future events the participant can vividly imagine as happening right now.
  Participants will be instructed to think about the EFT cues they created to help them focus on the future and importance of reaching their weight-loss goals. Participants will be instructed to use their EFT cues at least once per day, but will be encouraged to use their cues with every eating and physical activity decision.

SUMMARY:
Family-based treatments (FBT) for obesity have been shown to be effective in achieving significant weight reductionin overweight or obese children and parents [Altman & Wilfley, 2015]. One component of the current FBT programused in this study that has received little attention is thought training, specifically episodic future thinking (EFT). EFTteaches individuals to pre-experience events, or think prospectively, about future events as if they were happeningnow and has been shown to reduce delay discounting (DD) which is defined as discounting smaller rewards now for a larger reward in the [Daniel, Said, Stanton, & Epstein]. Furthermore, EFT has been shown to help people purchase fewer calories when they are grocery shopping [Hollis-Hansen et al., 2019], thereby displaying potential to be an effective measure in modulating the food environment in homes and may play a role in changing eating behaviors related to weight loss [Appelhaus et al.,2019].

Given the power of EFT in promoting the purchase of fewer calories, it is plausible that EFT training focused around grocery shopping during FBT could help shift one's thought processes towards healthier food choices, promoting behavioral change that has lasting impact on the home environment. Thus, the primary purpose of this study is to assess whether EFT training promotes active behavioral change pertaining to grocery shopping during FBT. In turn,this resulting behavior change could lead to healthier eating behavior and may promote weight loss for the whole family.

We hypothesize:

* There will be a reduction in BMI for adults/percent over BMI for children and weight from baseline
* There will be a reduction in delay discounting for children

DETAILED DESCRIPTION:
The study program is organized into 15 sessions. There is a mix of group sessions, individual family in-person sessions, and individual family phone sessions. Each session is outlined below:

WEEK 0 - Baseline Session: In-Lab Group Session - All Baseline sessions were completed as planned in lab.

First, upon arriving to the lab, each dyad will be escorted to a private room and will complete the following:

1. Have height and weight measured.
2. Complete surveys: Consideration of Future Consequences Scale (CFCS), EDE-Q (Parent), KEDS (Child)
3. Complete the Delay Discounting Task, the Online Grocery Shopping Task, and Home Food Inventory. A letter was sent to each family explaining the change from in-home visits with the Cupboard inventory to the self-completed Home Food Inventory, due to growing concern over COVID-19.
4. Receive first assessment payment ($40 dollars)

Following steps 1-4, the families will take part in a group session to learn the core components of the program in presentations by the research staff.

Weeks 1-14 ~ 1 hour; Weekly In-Lab Group Sessions - Due to the COVID 19 outbreak, in-person assessments and interventions are no longer feasible. Therefore, the researchers will carry out these study components remotely. The programs that will be used are phone, Zoom, and Qualtrics.

1. The day of their assigned parent group session, each family will email the study coordinator a photocopy of their food receipts, receipt forms, and food log. They will self-report weights via email as well.
2. Children will join a child-only Zoom group video session, and parents will join a parent-only Zoom video session. Each group will be led by a study team member. In these sessions, participants will do the thought training program, and talk to staff and other group members about progress in the program. Each parent-child dyad will meet via Zoom or phone at a separate time with a study team member to complete the case management portion of the program.

   1. During the 15-week intervention, participants will be asked to log their activity related to the program in food logs.
   2. Researchers will access the information and send feedback to the participants (via text, phone, and/or email) to help them succeed in the program.

Throughout the baseline period, the study team will assess all participants' adherence levels through looking at data from the food logs and the collected receipts.

Once a family has been determined to be adhering to the study protocol, the participant will then be randomly assigned to either the 7- week or 10-week baseline group. After the assigned baseline, participants will be eligible to start the EFT intervention.

An assessment session will take place the week the group starts the intervention, which will consist of 1- Self-reported weights via email 2- Complete surveys: EDE-Q (Parent), KEDS (Child) on Qualtrics 3- Complete EFT cue generation needed for thought training 4- Complete the Delay Discounting Task on Qualtrics and the Virtual Shopping Task via emailed instructions.

5- Review weekly receipts 6- Receive assessment session payment 7. Receive a EFT Cue Retrieval technology tutorial via emailed instructions, or a Zoom or phone session as requested

EFT Cue Retrieval: The experimenter will then train participants in both groups on how to retrieve cues from their cell phone or alternative WiFi device, to pay attention to and think about the cues, and how to adhere to the study's expectations for utilizing to the cues. Participants will be told to use their cues any time they need to, especially around eating episodes, using the prompt response website - Mobile Audio Management and Response Tracker (MAMRT)(Sze, Daniel, Kilanowski, Collins, Epstein, 2015).

Assessment measures must be completed the day of their assigned group sessions. Child and Parent Zoom-based group sessions will be conducted at their scheduled times, as well as scheduled case management.

Week 15 ~ Final Assessment - All assessment measures for week 15 will be conducted remotely, unless COVID-19related restrictions are lifted, in which an in-lab visit for final measurements may be conducted.

1. Self-reported heights and weights
2. Complete surveys on Qualtrics: Consideration of Future Consequences Scale (CFCS), EDE-Q (Parent), KEDS (Child),Formative Questionnaire, TT Frequency of Use
3. Complete the Delay Discounting Task, Shelf Life Inventory, and Home Food Inventory on Qualtrics, and the Virtual Shopping Task via emailed instructions.
4. Review weekly receipts and receive payment if applicable ($25 dollars) via check request, Amazon Pay or Forte.
5. Receive final assessment session payment ($45 dollars) via check request, Amazon Pay or Forte.

Assessment measures must be completed the day of their assigned group sessions. Child and Parent Zoom-based group sessions will be conducted at their scheduled times, as well as scheduled case management.

ELIGIBILITY:
Inclusion:

* Child age between 10-14
* Child height and weight that calculates to a BMI above the 85th percentile (BMI in overweight/obesity range)
* Parent height and weight that calculates to a BMI above 18
* Possession of at least one electronic device (per family) with WiFi capabilities (e.g. smartphone, tablet, computer)
* Home internet access
* Motivation to lose weight

Exclusion:

* Disordered eating patterns (e.g. binge-eating disorder, extreme weight-loss behaviors)
* A family history of eating disorders (siblings, children, parents, or grandparents)
* Medical conditions that are known to interfere with weight-loss (e.g. type 1 diabetes, thyroid disease)
* Medical conditions that may affect their ability to use the computer for a prolonged period of time or follow study protocol
* Psychopathology or disabilities that would limit adherence to protocol (e.g. depression, suicidality, ADHD). Participant will only be excluded if the disability would not allow them to adhere to protocol. Just having the disability does not exclude them. Suicidality would be automatically be exclusionary)
* Substance use, abuse, or dependence (e.g. binge drinkers, illicit substance users, alcoholics)
* Plans to start or stop a medication that may affect appetite/weight-loss during the intervention period
* Have started a medication within 6 months that is affecting appetite/weight-loss
* Plans to move out of the area during the treatment period
* Pregnancy/breastfeeding or plans of becoming pregnant during the study period
* Is participating in another weight-loss program
* Can not successfully record eating behavior in the MyFitnessPal app
* A) Had bariatric surgery less than one year ago B) If the potential participant had bariatric surgery over a year ago, their weight has not been stable for at least 6 months

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Epstein, PhD, Principal Investigator — State University of New York at Buffalo; Denise Wilfley, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daniel TO, Stanton CM, Epstein LH. The future is now: comparing the effect of episodic future thinking on impulsivity in lean and obese individuals. Appetite. 2013 Dec;71:120-5. doi: 10.1016/j.appet.2013.07.010. Epub 2013 Jul 31. PMID 23917063
- [Background] Benoit RG, Gilbert SJ, Burgess PW. A neural mechanism mediating the impact of episodic prospection on farsighted decisions. J Neurosci. 2011 May 4;31(18):6771-9. doi: 10.1523/JNEUROSCI.6559-10.2011. PMID 21543607
- [Background] Boyer P. Evolutionary economics of mental time travel? Trends Cogn Sci. 2008 Jun;12(6):219-24. doi: 10.1016/j.tics.2008.03.003. Epub 2008 May 28. PMID 18468941
- [Background] Daniel TO, Said M, Stanton CM, Epstein LH. Episodic future thinking reduces delay discounting and energy intake in children. Eat Behav. 2015 Aug;18:20-4. doi: 10.1016/j.eatbeh.2015.03.006. Epub 2015 Mar 28. PMID 25863227
- [Background] Atance CM, O'Neill DK. Episodic future thinking. Trends Cogn Sci. 2001 Dec 1;5(12):533-539. doi: 10.1016/s1364-6613(00)01804-0. PMID 11728911
- [Background] John LK, Loewenstein G, Troxel AB, Norton L, Fassbender JE, Volpp KG. Financial incentives for extended weight loss: a randomized, controlled trial. J Gen Intern Med. 2011 Jun;26(6):621-6. doi: 10.1007/s11606-010-1628-y. Epub 2011 Jan 20. PMID 21249462
- [Background] Leahey TM, Fava JL, Seiden A, Fernandes D, Doyle C, Kent K, La Rue M, Mitchell M, Wing RR. A randomized controlled trial testing an Internet delivered cost-benefit approach to weight loss maintenance. Prev Med. 2016 Nov;92:51-57. doi: 10.1016/j.ypmed.2016.04.013. Epub 2016 Apr 17. PMID 27095323

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Particpants were parent-child dyads, so each unit dyad consists of 1 parent and 1 child, e.g. 4 dyads enrolled in Episodic future thinking group 7-week baseline and 3 dyads enrolled in episodic future thinking group 10-week baseline
Groups:
- Episodic Future Thinking Group 7-week Baseline: The experimental group will receive the Episodic Future Thinking (EFT) intervention after a 7-week baseline.
  EFT teaches individuals to pre-experience events, or think prospectively, about future events as if they were happening now [Atance].
  Episodic Future Thinking Group: Participants in the Episodic Future Thinking (EFT) Group will train with EFT throughout the entire study. As part of the training, research staff will help participants create "cues." Cues are descriptions of future events the participant can vividly imagine as happening right now.
  Participants will be instructed to think about the EFT cues they created to help them focus on the future and importance of reaching their weight-loss goals. Participants will be instructed to use their EFT cues at least once per day, but will be encouraged to use their cues with every eating and physical activity decision.
- Episodic Future Thinking Group 10-week Baseline: The experimental group will receive the Episodic Future Thinking (EFT) intervention after a 10-week baseline.
  EFT teaches individuals to pre-experience events, or think prospectively, about future events as if they were happening now [Atance].
  Episodic Future Thinking Group: Participants in the Episodic Future Thinking (EFT) Group will train with EFT throughout the entire study. As part of the training, research staff will help participants create "cues." Cues are descriptions of future events the participant can vividly imagine as happening right now.
  Participants will be instructed to think about the EFT cues they created to help them focus on the future and importance of reaching their weight-loss goals. Participants will be instructed to use their EFT cues at least once per day, but will be encouraged to use their cues with every eating and physical activity decision.
Period: Overall Study
Arm/Group | Episodic Future Thinking Group 7-week Baseline | Episodic Future Thinking Group 10-week Baseline
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline participants included 7 parent-child dyads. Baseline characteristics are broken down by parent and child information on separate lines.
Groups:
- Total: Total of all reporting groups
Arm/Group | Episodic Future Thinking Group 7-week Baseline | Episodic Future Thinking Group 10-week Baseline | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] — Parent age, years Population: Parent information n = 7
  years | 39.5 (6.9) | 38.0 (7.2) | 38.9 (6.5)
Age, Continuous [Mean (Standard Deviation); unit: years] — Child Age, years Population: child information n = 7
  years | 10.5 (0.6) | 10.7 (0.6) | 10.6 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Parent reported sex Population: Parent information n = 7
  Participants
    Female | 4 | 3 | 7
    Male | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Child reported Sex Population: child information n = 7
  Participants
    Female | 2 | 2 | 4
    Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Parent self-reported Ethnicity Population: Parent information n = 7
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 4 | 3 | 7
    Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Child self-reported ethnicity Population: child information n = 7
  Participants
    Hispanic or Latino | 1 | 0 | 1
    Not Hispanic or Latino | 3 | 3 | 6
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Parent self-reported Race Population: Parent information n = 7
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 1 | 1
    White | 3 | 2 | 5
    More than one race | 1 | 0 | 1
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Child self-reported race Population: child information n = 7
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 1 | 2
    White | 3 | 2 | 5
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: dyads]
  United States | 4 | 3 | 7
Parent Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Parent body mass index as calculated BMI = kg/m^2. Overweight is defined for adults as BMI<30 and BMI>=25 and obesity as BMI>=30 Population: Parent BMI is reported (n = 7)
  kg/m^2 | 32.7 (16.8) | 36.9 (7.9) | 34.5 (12.9)
Child BMI percentile [Mean (Standard Deviation); unit: standardized percentile] — BMI percentile is used for children rather than BMI, as it is standardized for child age and sex. BMI percentile >=95th is considered obesity for children and BMI>=85 and <95th is considered overweight for children Population: Child (n = 7) measured BMI percentile
  standardized percentile | 95.5 (4.7) | 95.7 (3.1) | 95.6 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in BMI for Parent Participants From Baseline at Weeks 8, 11 and 15
Description: Height (cm) and weight (lbs) will be assessed to calculate BMI (kg/m^2) for parents. Change will be assessed at baseline, week 8, 11 and 15 from baseline.
Time Frame: Change from Baseline BMI at week 8, 11 and 15
Population: Parents (n = 7) will be analyzed for change in BMI from baseline
Measure: Mean (Standard Deviation); unit: kg/m^2
Groups:
- Episodic Future Thinking Group 7-week Baseline: The experimental group will receive the Episodic Future Thinking (EFT) intervention after 7-weeks. EFT teaches individuals to pre-experience events, or think prospectively, about future events as if they were happening now [Atance].
  Episodic Future Thinking Group: Participants in the Episodic Future Thinking (EFT) Group will train with EFT throughout the entire study. As part of the training, research staff will help participants create "cues." Cues are descriptions of future events the participant can vividly imagine as happening right now.
  Participants will be instructed to think about the EFT cues they created to help them focus on the future and importance of reaching their weight-loss goals. Participants will be instructed to use their EFT cues at least once per day, but will be encouraged to use their cues with every eating and physical activity decision.
- Episodic Future Thinking 10-week Baseline: The experimental group will receive the Episodic Future Thinking (EFT) intervention after 10-weeks. EFT teaches individuals to pre-experience events, or think prospectively, about future events as if they were happening now [Atance].
  Episodic Future Thinking Group: Participants in the Episodic Future Thinking (EFT) Group will train with EFT throughout the entire study. As part of the training, research staff will help participants create "cues." Cues are descriptions of future events the participant can vividly imagine as happening right now.
  Participants will be instructed to think about the EFT cues they created to help them focus on the future and importance of reaching their weight-loss goals. Participants will be instructed to use their EFT cues at least once per day, but will be encouraged to use their cues with every eating and physical activity decision.
Arm/Group | Episodic Future Thinking Group 7-week Baseline | Episodic Future Thinking 10-week Baseline
Number analyzed (Participants) | 4 | 3
kg/m^2
  Parent Baseline BMI | 32.7 (16.8) | 36.9 (7.9)
  Change in parent BMI from baseline to week 8 | -1.3 (1.2) | -1.9 (1.0)
  Change in Parent BMI from baseline to week 11 | -1.7 (1.2) | -2.2 (0.9)
  Change in parent BMI from baseline to week 15 | -1.9 (1.6) | -2.6 (0.9)
Statistical Analysis 1: Comparison: Episodic Future Thinking Group 7-week Baseline vs Episodic Future Thinking 10-week Baseline; Change in parent BMI from baseline at 8,11 to 15 weeks; Test type: Superiority; p < 0.01, ANOVA; Mean Difference (Net) = 2.2 — This mean difference represents the main effect of time from baseline to 15 weeks, regardless of group

2. Primary Outcome: Change in Weight for Parents From Baseline at Weeks 8, 11 and 15
Description: Weight was measured in lbs
Time Frame: Change from Baseline weight at week 8, 11 and 15
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Episodic Future Thinking Group 7-week Baseline | Episodic Future Thinking Group 10-week Baseline
Number analyzed (Participants) | 4 | 3
pounds
  Change in weight (lbs) from 0 to 8 weeks | -5.8 (2.6) | -7.2 (3.0)
  Change in weight (lbs) from 0 to 11 weeks | -8.5 (2.4) | -9.1 (2.1)
  Change in weight (lbs) from 0 to 15 weeks | -9.6 (5.1) | -11.7 (2.7)
Statistical Analysis 1: Comparison: Episodic Future Thinking Group 7-week Baseline; repeated measures analysis of variance for time (0,8,11,15 weeks) for weight change (lbs); Test type: Superiority; p = 0.003, ANOVA — main effect of time; Mean Difference (Net) = -10.5 — This is the main effect of weight change at week 15, e.g. average weight change from baseline to week 15 in the entire sample of parents

3. Primary Outcome: Change in BMI Percentile for Children
Description: Change in BMI percentile for children from 0, 8, 11 and 15 weeks
Time Frame: Baseline, 8, 11 and 15 weeks
Population: Children (n = 7) analysis
Measure: Mean (Standard Deviation); unit: Standardized percentile
Groups:
- Episodic Future Thinking 10-week Baseline: The experimental group will receive the Episodic Future Thinking (EFT) intervention after a 10-week baseline. EFT teaches individuals to pre-experience events, or think prospectively, about future events as if they were happening now [Atance].
  Episodic Future Thinking Group: Participants in the Episodic Future Thinking (EFT) Group will train with EFT throughout the entire study. As part of the training, research staff will help participants create "cues." Cues are descriptions of future events the participant can vividly imagine as happening right now.
  Participants will be instructed to think about the EFT cues they created to help them focus on the future and importance of reaching their weight-loss goals. Participants will be instructed to use their EFT cues at least once per day, but will be encouraged to use their cues with every eating and physical activity decision.
Arm/Group | Episodic Future Thinking Group 7-week Baseline | Episodic Future Thinking 10-week Baseline
Number analyzed (Participants) | 4 | 3
Standardized percentile
  Baseline Child BMI percentile | 95.5 (4.8) | 95.7 (3.1)
  Change in child BMI percentile from baseline to 8 weeks | -1.8 (2.8) | -4.3 (5.9)
  change in child BMI percentile from 0 to 11 weeks | -1.7 (2.9) | -4.9 (6.4)
  Change in child BMI percentile from baseline to 15 weeks | -1.3 (3.9) | -4.3 (4.5)
Statistical Analysis 1: Comparison: Episodic Future Thinking Group 7-week Baseline; Repeated measures ANOVA for child BMI percentile at 0, 8, 11 and 15 weeks; Test type: Superiority; p = 0.06, ANOVA; Mean Difference (Final Values) = -2.6 — average difference in BMI percentile for entire sample

4. Secondary Outcome: Delay Discounting for Children
Description: Delay Discounting will be measured using monetary Delay Discounting tasks with $100 as the delayed reward. Delay discounting is assessed using Area Under the Curve (AUC), or time*indifference point/delay. AUC for delay discounting included time (x-axis) and indifference point (y-axis), or the amount of money at which the immediate and delayed options are approximately equal. Indifference points are a proportion of the max amount (range 0 - 100) and delays are calculated as proportion of max delay. AUC adds the calculated areas for each timepoint from the previous timepoint. AUC ranges from 0 (most impulsive, did not choose delay) to 100 (least impulsive, always chose delay). As this is a measure that is standardized, units are proportion of maximum delayed reward x proportion of maximum delay.
Time Frame: Baseline, 10 weeks, 15 weeks
Population: n = 7 children
Measure: Mean (Standard Deviation); unit: proportion max reward x proportion delay
Arm/Group | Episodic Future Thinking Group 7-week Baseline | Episodic Future Thinking 10-week Baseline
Number analyzed (Participants) | 4 | 3
proportion max reward x proportion delay
  Baseline Area Under the curve | 0.28 (0.13) | 0.22 (0.06)
  Week 10 Area under the curve | 0.34 (0.17) | 0.35 (0.15)
  Week 15 Area under the curve | 0.36 (0.12) | 0.35 (0.14)
Statistical Analysis 1: Comparison: Episodic Future Thinking Group 7-week Baseline vs Episodic Future Thinking 10-week Baseline; repeated measures ANOVA, reporting repeated measures effect only; Test type: Superiority; p = 0.07, ANOVA; Mean Difference (Final Values) = 0.10 — average change in delay discounting measure area under the curve for all participants (parents and children) in both groups from baseline to week 15

5. Primary Outcome: Change in Weight for Children From Baseline at Weeks 8, 11 and 15
Description: Weight was measured in lbs and examined as change from baseline in lbs at week 8, 11 and 15
Time Frame: Change from Baseline weight at week 8, 11 and 15
Population: child
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Episodic Future Thinking Group 7-week Baseline | Episodic Future Thinking Group 10-week Baseline
Number analyzed (Participants) | 4 | 3
pounds
  Change in weight (lbs) from 0 to 8 weeks | -0.78 (2.61) | -2.50 (4.30)
  Change in weight (lbs) from 0 to 11 weeks | -0.73 (3.20) | -1.73 (6.23)
  Change in weight (lbs) from 0 to 15 weeks | -0.08 (4.41) | -1.77 (4.85)
Statistical Analysis 1: Comparison: Episodic Future Thinking Group 7-week Baseline vs Episodic Future Thinking Group 10-week Baseline; Test type: Superiority; p = 0.64, ANOVA; Mean Difference (Net) = -0.8 — Difference between weight at baseline and week 15 in lbs for all children, regardless of group

ADVERSE EVENTS:
Time Frame: 15 weeks during which families received treatment
Groups:
- Episodic Future Thinking Group - 7 Week Parents: Parent participants of the family dyad.
  The experimental group will receive the Episodic Future Thinking (EFT) intervention after a 7-week baseline. EFT teaches individuals to pre-experience events, or think prospectively, about future events as if they were happening now [Atance].
  Episodic Future Thinking Group: Participants in the Episodic Future Thinking (EFT) Group will train with EFT throughout the entire study. As part of the training, research staff will help participants create "cues." Cues are descriptions of future events the participant can vividly imagine as happening right now.
  Participants will be instructed to think about the EFT cues they created to help them focus on the future and importance of reaching their weight-loss goals. Participants will be instructed to use their EFT cues at least once per day, but will be encouraged to use their cues with every eating and physical activity decision.
- Episodic Future Thinking Group 7-week Children: Child participants of the family dyad.
  The experimental group will receive the Episodic Future Thinking (EFT) intervention after a 7-week baseline. EFT teaches individuals to pre-experience events, or think prospectively, about future events as if they were happening now [Atance].
  Episodic Future Thinking Group: Participants in the Episodic Future Thinking (EFT) Group will train with EFT throughout the entire study. As part of the training, research staff will help participants create "cues." Cues are descriptions of future events the participant can vividly imagine as happening right now.
  Participants will be instructed to think about the EFT cues they created to help them focus on the future and importance of reaching their weight-loss goals. Participants will be instructed to use their EFT cues at least once per day, but will be encouraged to use their cues with every eating and physical activity decision.
- Episodic Future Thinking Group - 10 Week Parents: Parent participants of the family dyad.
  The experimental group will receive the Episodic Future Thinking (EFT) intervention after a 10-week baseline. EFT teaches individuals to pre-experience events, or think prospectively, about future events as if they were happening now [Atance].
  Episodic Future Thinking Group: Participants in the Episodic Future Thinking (EFT) Group will train with EFT throughout the entire study. As part of the training, research staff will help participants create "cues." Cues are descriptions of future events the participant can vividly imagine as happening right now.
  Participants will be instructed to think about the EFT cues they created to help them focus on the future and importance of reaching their weight-loss goals. Participants will be instructed to use their EFT cues at least once per day, but will be encouraged to use their cues with every eating and physical activity decision.
- Episodic Future Thinking Group - 10 Week Children: Child participants of the family dyad.
  The experimental group will receive the Episodic Future Thinking (EFT) intervention after a 10-week baseline. EFT teaches individuals to pre-experience events, or think prospectively, about future events as if they were happening now [Atance].
  Episodic Future Thinking Group: Participants in the Episodic Future Thinking (EFT) Group will train with EFT throughout the entire study. As part of the training, research staff will help participants create "cues." Cues are descriptions of future events the participant can vividly imagine as happening right now.
  Participants will be instructed to think about the EFT cues they created to help them focus on the future and importance of reaching their weight-loss goals. Participants will be instructed to use their EFT cues at least once per day, but will be encouraged to use their cues with every eating and physical activity decision.
Arm/Group | Episodic Future Thinking Group - 7 Week Parents | Episodic Future Thinking Group 7-week Children | Episodic Future Thinking Group - 10 Week Parents | Episodic Future Thinking Group - 10 Week Children
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/25/NCT03731325/Prot_SAP_000.pdf